CLINICAL TRIAL: NCT00830531
Title: Pilot Study of Bumetanide for Newborn Seizures: A Phase I Study of Pharmacokinetics and Safety of Bumetanide for Neonatal Seizures
Brief Title: Pilot Study of Bumetanide for Newborn Seizures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soul, Janet , M.D. (Individual)
Collaborators: Citizens United for Research in Epilepsy (Other); Harvard Catalyst- Harvard Clinical and Translational Science Center (Unknown); Translational Research Program, Boston Children's Hospital (Unknown); Charles H. Hood Foundation (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Mooney Family Initiative for Translational Studies in Rare Diseases, Boston Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CURE 07120492; 1R01NS066929-01A1 (NIH)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Seizures
Keywords: Hypoxic-ischemic encephalopathy; Neonatal stroke; Intracranial hemorrhage; Perinatal asphyxia; Neonatal Seizures
MeSH Terms: conditions — Seizures; Hypoxia-Ischemia, Brain; Intracranial Hemorrhages | interventions — Bumetanide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Standard phenobarbital combined with either 0.1 mg/kg, 0.2 mg/kg, or 0.3 mg/kg of bumetanide as determined by the status of the dose escalation design.
  Interventions: Drug: Bumetanide
- 2 (Placebo Comparator): Standard phenobarbital therapy combined with normal saline as placebo for bumetanide
  Interventions: Drug: Normal Saline as Placebo

INTERVENTIONS:
Drug: Bumetanide — Bumetanide either 0.1 mg/kg, 0.2 mg/kg or 0.3 mg/kg IV administered together with standard phenobarbital therapy
  Other Names: Bumex
  Arms: 1
Drug: Normal Saline as Placebo — Normal Saline as placebo for bumetanide either 0.1 mg/kg, 0.2 mg/kg or 0.3 mg/kg IV administered together with standard phenobarbital therapy
  Other Names: 0.9% NaCl
  Arms: 2

SUMMARY:
The main goal of the study is to obtain pharmacokinetic and safety data of bumetanide in newborns with refractory seizures. The overall hypothesis is that bumetanide, added to conventional antiepileptic (antiseizure) medications, will be a safe and well tolerated medication, compared with conventional antiepileptic drugs alone.

DETAILED DESCRIPTION:
Seizures occur more often during the newborn period (2-3.5 per 1000 live births) than at any later age. Neonatal seizures can lead to frequent and serious long-term consequences in survivors, such as later epilepsy and significant cognitive and motor disabilities. Unfortunately there are no completely effective drugs to treat neonatal seizures. Anti-epileptic drugs (AEDs) currently used to treat neonatal seizures are generally ineffective and have significant potential for side effects. Furthermore, many of these AEDs have never been tested in a randomized study. Numerous experts have thus emphasized in the last few years the urgent need for randomized trials of potential new treatments for neonatal seizures. The investigators are conducting a pilot study of the drug bumetanide as one such potential and novel treatment. Bumetanide is a commercially available drug that has been used safely in newborns as a diuretic for many years with minimal side effects. Recent basic science research in animals has shown bumetanide to be very effective in reducing seizures in neonatal animals by blocking a specific chloride importer which is highly expressed in neonates but not in children and adults (1). Moreover, these experimental studies have shown bumetanide to be particularly effective against seizures when used in combination with phenobarbital (PB), which is the standard first drug given to treat neonatal seizures (2).

The investigators will conduct a randomized, double-blind, controlled, dose escalation study of BTN as add-on therapy to treat refractory seizures caused by HIE, focal or multi-focal stroke, intracranial hemorrhage, CNS infection, genetic syndrome, focal or diffuse brain malformation, idiopathic or presumed genetic etiology of seizures, or metabolic disorder other than electrolyte disturbances or those caused by renal failure not controlled by an initial loading dose of PB. The trial will test the feasibility of early enrollment of newborns with HIE, rapid application of a full montage EEG, and continuous review of EEG data to detect refractory seizures as soon as they occur following an initial loading dose of PB. When an EEG-proven seizure occurs at least 30 minutes following a loading dose of PB, the newborn will be randomized to receive either BTN or placebo in conjunction with a loading dose of PB. Clinical, laboratory and continuous EEG monitoring data obtained after BTN administration will be analyzed to determine the pharmacokinetics (3) and safety of BTN by comparing data from treatment and standard therapy groups. This study addresses important challenges in trial design and sets the stage for trials to improve treatment of neonatal seizures. Data from this pilot study will be used to guide design of a planned Phase III multicenter trial to test the efficacy of BTN to control refractory neonatal seizures.

ELIGIBILITY:
Inclusion Criteria:

* newborns with a post-conceptional age of 33-44 weeks
* condition with risk for seizure:

  * asphyxia
  * intracranial hemorrhage
  * suspected or confirmed stroke
  * CNS infection
  * genetic syndrome
  * focal or diffuse brain malformation
  * idiopathic or presumed genetic etiology of seizures
  * metabolic disorder other than electrolyte disturbances or those caused by renal failure
* suspected clinical seizure

Exclusion Criteria:

* have transient metabolic abnormalities (e.g., transient hypocalcemia) as the sole cause of seizures
* are receiving ECMO (extracorporeal membrane oxygenation) therapy because of alteration of bumetanide pharmacokinetics by ECMO
* have contraindications to bumetanide (as determined by treating physician)
* have received diuretics such as furosemide or BTN
* newborns with a total serum bilirubin > 15 mg/dL at enrollment
* newborns given ≥ 40mg/kg of phenobarbital
* loading doses of AEDs other than phenobarbital (those who receive levetiracetam are still eligible since levetiracetam does not affect bumetanide pharmacokinetics)

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2010-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is determination of the pharmacokinetics and safety of bumetanide in newborns with refractory seizures. | 6-7 years are anticipated for the collection of the neonatal data
  The investigators will determine the dose exposure, half-life, volume of distribution and clearance of bumetanide in newborns with refractory seizures. The investigators will determine if there is a significant effect of hepatic dysfunction or hypothermia on bumetanide pharmacokinetics. For evaluation of safety, the rate of adverse events will be compared between treatment and control groups.

SECONDARY OUTCOMES:
A secondary outcome is determination of the feasibility of the study design to test antiepileptic drugs to treat neonatal seizures caused by acute hypoxic-ischemic encephalopathy in a clinical trial. | 6-7 years are anticipated for collection of the neonatal data
  The investigators will determine the feasibility of enrolling and randomizing newborns early in the course of their refractory seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Soul, MD,CM, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (4):
  - Tufts Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Dzhala VI, Talos DM, Sdrulla DA, Brumback AC, Mathews GC, Benke TA, Delpire E, Jensen FE, Staley KJ. NKCC1 transporter facilitates seizures in the developing brain. Nat Med. 2005 Nov;11(11):1205-13. doi: 10.1038/nm1301. Epub 2005 Oct 9. PMID 16227993
- [Background] Dzhala VI, Brumback AC, Staley KJ. Bumetanide enhances phenobarbital efficacy in a neonatal seizure model. Ann Neurol. 2008 Feb;63(2):222-35. doi: 10.1002/ana.21229. PMID 17918265
- [Background] Li Y, Cleary R, Kellogg M, Soul JS, Berry GT, Jensen FE. Sensitive isotope dilution liquid chromatography/tandem mass spectrometry method for quantitative analysis of bumetanide in serum and brain tissue. J Chromatogr B Analyt Technol Biomed Life Sci. 2011 Apr 15;879(13-14):998-1002. doi: 10.1016/j.jchromb.2011.02.018. Epub 2011 Feb 19. PMID 21414852
- See also: Publication reporting bumetanide trial results, Annals of Neurology 2020 — https://pubmed.ncbi.nlm.nih.gov/33201535/